CLINICAL TRIAL: NCT07251413
Title: Phase Ib/II Study Of The Combination Of Cemiplimab Plus Imiquimod and Laser Therapy As Neoadjuvant Treatment In Cutaneous Basal Cell Carcinoma
Brief Title: Cemiplimab Plus Imiquimod and Laser Therapy As Neoadjuvant Treatment In Cutaneous Basal Cell Carcinoma
Acronym: CEMIQUID
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto Oncológico Dr Rosell (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOR-REG-2501; 2025-520698-38-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-29; First posted 2025-11-26 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Cutaneous Basal Cell Carcinoma
Keywords: Cutaneous Carcinoma; Cemiplimab; Imiquimod; Laser Therapy
MeSH Terms: interventions — cemiplimab; Imiquimod

STUDY DESIGN:
Intervention Model Description: CEMIQUID is a multi-center, open-label, phase Ib/II, two-cohort study for patients with high risk, potentially resectable basal cell carcinoma (BCC). Patients enrolled in the Phase II part of the study will be randomly assigned to Cemiplimab +/- Imiquimod
  The study is divided into two phases:
  Phase Ib: 6 patients will be included and the main objective will be to evaluate the safety and toxicity of the combination of intravenous cemiplimab plus topical imiquimod (plus fractional laser therapy) as neoadjuvant treatment in patients with high risk and potentially resectable BCC.
  Phase II: If the treatment is deemed feasible on Phase Ib, 12 additional patients will be included to evaluate the antitumoral activity in terms of 3-years rate of relapse-free survival (RFS) according to RECIST 1.1 (Appendix 3) of intravenous cemiplimab as single therapy or in combination with topical imiquimod (plus fractional laser therapy) as neoadjuvant treatment in patients with high risk and potentially re
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: cemiplimab neoadjuvant treatment (Active Comparator): Patients will be treated with single agent intravenous cemiplimab 350 mg every 3 weeks for a total of 4 neoadjuvant cycles (12 weeks).
  Interventions: Drug: cemiplimab
- Cohort 2: cemiplimab plus topical imiquimod (plus fractional laser therapy) as neoadjuvant (Experimental): Patients will be treated with intravenous cemiplimab 350 mg every 3 weeks in combination with topical imiquimod 5% cream self-applied once daily 5 days per week (plus low-intensity laser therapy at 1- or 3-week interval), for a total of 4 neoadjuvant cycles (12 weeks).
  Interventions: Drug: cemiplimab; Drug: Topical imiquimod

INTERVENTIONS:
Drug: cemiplimab — cemiplimab 350 mg every 3 weeks for a total of 4 neoadjuvant cycles (12 weeks).
Drug: Topical imiquimod — Topical imiquimod 5% cream self-applied once daily 5 days per week (plus low-intensity laser therapy at 1- or 3-week interval),
  Arms: Cohort 2: cemiplimab plus topical imiquimod (plus fractional laser therapy) as neoadjuvant

SUMMARY:
Basal cutaneous cell carcinoma (BCC) is the most common skin cancer. Early-stage disease is managed with surgery or radiation that cure more than 95% of patients. Surgical excision is the treatment of choice and by far the most convenient and effective means of achieving cure of any invasive BCC, Surgery is rarely contra-indicated even in old, debilitated patients, but in locally advanced tumors surgery has the potential of having functional and cosmetic consequences, due to a big tumor size or difficult locations and it is not uncommon tumors that are borderline for the indication of curative surgery. Patients with high-risk disease who have large primary lesions are usually not amenable to a definitive cure with local intervention and may experience significant morbidity, disfigurement, or functional deficits. In some patients, the tumors recur and progress locally being radiotherapy and Hedgehog inhibition therapy available options.

Recently, cemiplimab was the first immunotherapy approved by the FDA and EMEA for locally advanced BCC after Hedgehog pathway inhibition The imiquimod (1-(2-methylpropyl)-1-H-imidazole [4,5-c] quinolone-amine) is a synthetic compound capable of activating the cells of the immune system, helping to control viruses, tumors, and intracellular parasites The combination of imiquimod plus anti PD-1 antibody could be synergistic.

The main hypoteis is that combining cemiplimab, an immune checkpoint inhibitor targeting PD-1, and local treatment with the Toll-like receptor 7 (TLR7) agonist imiquimod may increase immune response against tumor and result in an increase in the rate of definitive cure y in patients with basal cell carcinoma (BCC) who have a high risk of recurrence after surgery alone or a high risk of morbidity, disfigurement, or functional deficits: to increase the rate of definitive cure.

The CEMIQUID study main aims to evaluate:

1. The safety and toxicity of the combination of intravenous cemiplimab plus topical imiquimod (plus fractional laser therapy) as neoadjuvant treatment in patients with high risk and potentially resectable BCC.
2. The antitumoral activity in terms of 3-years rate of relapse-free survival (RFS) according to RECIST 1.1 of intravenous cemiplimab as single therapy or in combination with topical imiquimod plus fractional laser therapy as neoadjuvant treatment in patients with high risk and potentially resectable BCC.

Patients with high risk, potentially resectable basal cell carcinoma (BCC), enrolled in the Phase Ib part of the study will receive treatment with intravenous (iv) cemiplimab plus topical imiquimod plus fractional laser therapy as neoadjuvant treatment.

Patients enrolled in the Phase II part will be randomized to receive neoadjuvant cemiplimab as a single agent or the Phase Ib combination with imiquimod and fractional laser therapy

DETAILED DESCRIPTION:
1. RATIONALE Combining cemiplimab, an immune checkpoint inhibitor targeting PD-1, and local treatment with the Toll-like receptor 7 (TLR7) agonist imiquimod may increase immune response against tumor and result in an increase in the rate of definitive cure y in patients with basal cell carcinoma (BCC) who have a high risk of recurrence after surgery alone or a high risk of morbidity, disfigurement, or functional deficits: to increase the rate of definitive cure.
2. OBJECTIVE Combining cemiplimab, an immune checkpoint inhibitor targeting PD-1, and local treatment with the Toll-like receptor 7 (TLR7) agonist imiquimod may increase immune response against tumor and result in an increase in the rate of definitive cure y in patients with basal cell carcinoma (BCC) who have a high risk of recurrence after surgery alone or a high risk of morbidity, disfigurement, or functional deficits: to increase the rate of definitive cure.

   Primary objective:
   * The primary objective for the Phase Ib part of the trial is to evaluate the safety and toxicity of the combination of intravenous cemiplimab plus topical imiquimod (plus fractional laser therapy) as neoadjuvant treatment in patients with high risk and potentially resectable BCC.
   * The primary objective for the Phase II of the trial it to evaluate the antitumoral activity in terms of 3-years rate of relapse-free survival (RFS) according to RECIST 1.1 of intravenous cemiplimab as single therapy or in combination with topical imiquimod (plus fractional laser therapy) as neoadjuvant treatment in patients with high risk and potentially resectable BCC.

   Secondary objectives:
   * To evaluate pathological complete response rate (pCR) according to Immune-Related Pathologic Response Criteria' (irPRC) criteria.
   * To evaluate the activity in terms of response rate (RECIST 1.1), duration of response, clinical benefit, RFS/PFS and OS.
   * To evaluate the rate of resectability (downstaging) of BCC after 4 cycles of treatment.
   * To evaluate safety of the intended treatment regimen based on the frequency and severity of adverse events and Treatment-related adverse events (TRAEs) assessed by NCI CTCAE v5.0.
   * Translational research
3. PRIMARY TRIAL ENDPOINTS

   * Phase Ib: incidence of adverse events (AE) and treatment-related AEs (TRAEs) assessed by NCI CTCAE v5.0
   * Phase II: RFS rate at 3 years, defined as the proportion of patients free of locoregional progression or recurrence, distant metastasis (RECIST v 1.1).
4. SECONDARY TRIAL ENDPOINTS

   * Pathologic complete response (pCR)
   * Objective response rate (ORR)
   * Clinical benefit rate (CBR)
   * Duration of clinical benefit (DBC)
   * Relapse-free survival (RFS)
   * Overall survival (OS)
   * Adverse events (AE) and treatment-related AEs (TRAEs)
   * Molecular alterations in biological samples
5. TRIAL DESIGN

   CEMIQUID is a multi-center, open-label, phase Ib/II, two-cohort study. The study is divided into two phases:

   Phase Ib: 6 patients will be included and the main objective will be to evaluate the safety and toxicity of the combination of intravenous cemiplimab plus topical imiquimod (plus fractional laser therapy) as neoadjuvant treatment in patients with high risk and potentially resectable BCC.

   Phase II: If the treatment is deemed feasible on Phase Ib, 12 additional patients will be included to evaluate the antitumoral activity.

   On treatment clinic visits will occur every 3 weeks ±3 days. Computed tomography (CT), digital photography and lymph node ultrasonography (if applicable) will be used at baseline, prior to the third dose of neoadjuvant cemiplimab and prior to surgery to assess tumor response. Long term follow up of tumor evolution after surgical intervention will adhere to local standard clinical practice. The trial includes the assessment of safety (AEs, comorbidities) throughout the study period at every visit, and an exploratory study to evaluate the prognostic value and correlation between clinical features or molecular alterations.
6. TRIAL POPULATION

   Patients with high risk, potentially resectable basal cell carcinoma (BCC). High risk is defined as any of the following:
   1. at least 1 large lesion still resectable, but with increased risk for cosmetic disfigurement or functional defects by assessment of the enrolling physician.
   2. Having basosquamous, infiltrative, sclerosing/morpheaform, micronodular, and BCC with carcinosarcomatous differentiation features.
   3. Patients with large (≥ 3 cm in diameter in areas of intermedium risk of recurrence such as forehead, cheek, chin, neck, scalp or ≥ 5 cm for lesions in trunk/extremities) recurrent BCC.
   4. Multicentric tumors that would require a cosmetic disfigurement or functional defects.
7. STUDY TREATMENT

   All patients enrolled in the Phase Ib part of the study will receive treatment with intravenous (iv) cemiplimab 350 mg every 3 weeks plus topical imiquimod 5% cream self-applied once daily 5 days per week, and ablative fractional CO2 laser 10.600nm (±10nm) at 1- or 3-week intervals, for a total of 4 neoadjuvant cycles (12 weeks). The study treatment may be discontinued prematurely in case of unacceptable toxic effects, or disease progression.

   Patients enrolled in the Phase II part will be randomized to receive neoadjuvant cemiplimab 350 mg every 3 weeks as a single agent or the Phase Ib combination with imiquimod and CO2 laser.
8. ETHICAL CONSIDERATION

Cemiplimab is approved and might be considered the standard of care for patients with metastatic or locally advanced BCC who are not candidates for curative surgery. Imiquimod is a topical standard treatment for patients with BCC. Patients with high risk BCC require surgeries that may involve comorbidities or disfigurement. Combining both treatments may have a synergistic activity and induce tumor size reduction easing its resection.

The neoadjuvant timings proposed will not substantially delay the surgical intervention. The use of 4 doses of cemiplimab in the neoadjuvant setting has been previously tested in 79 patients with CSCC and resulted in a feasible and safe therapy.

The study is designed as Ib because doses recommended for cemiplimab and imiquimod are well justified by previous experience in clinical trials and use under marketed conditions. Given the different mechanisms of action and the type of administration, it is not expected to have overlapping toxicities that may require dose modifications of the initial recommended doses. Therefore, dose escalation is not required and the trial includes the dosing of one or more cohorts of patients at the recommended dose. The potential risks of cemiplimab and imiquimod are well known based on clinical trials and marketing experience. Most frequent AEs are immune-related and could be properly managed with adequate care. The protocol already includes safety measures to minimize the risks.

Therefore, the potential benefits of cemiplimab and imiquimod as combined neoadjuvant treatmnt in patients with BCC outweigh the risks.

The study will be conducted in accordance with the principles of the Helsinki Declaration Adopted by the 18th World Medical Assembly, Helsinki, Finland, June 1964 updated to its latest version Helsinki, Finland, October 2024. With the Good Clinical Practice (GCP) standards issued by the Working Party on Medicinal Product Efficacy of the European Economic Community (1990) (CPMP / ICH / 135/95).

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent.
2. Histologically confirmed diagnosis of basal cell carcinoma (BCC), potentially resectable with curative intention.

   1. The definition of resectability will be determined locally by the surgeon according to his/her criteria and local standard guidelines. The validated classification from University Hospital of Lille should be used for guidance in resectability assessment (Appendix 11).
   2. Surgery would be recommended in routine clinical practice.
3. Patient should be considered as high risk, defined as:

   1. at least 1 large lesion (≥ 2 cm in diameter in trunk/extremities or any size in Head, neck, hands, feet, pretibial, and anogenital) still resectable, but with increased risk for cosmetic disfigurement or functional defects by assessment of the enrolling physician.
   2. Having basosquamous, infiltrative, sclerosing/morpheaform, micronodular, and BCC with carcinosarcomatous differentiation features in any portion of the tumor.
   3. Patients with large (≥ 3 cm in diameter in areas of intermedium risk of recurrence such as forehead, cheek, chin, neck, scalp or ≥ 5 cm for lesions in trunk/extremities) recurrent basal cell carcinoma are also eligible.
   4. Multicentric tumors that would require a cosmetic disfigurement or functional defects by assessment of the enrolling physician will be eligible.
4. At least one measurable lesion by RECIST v1.1 (Appendix 3).
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
6. Life expectancy of at least 24 weeks.
7. Pretreatment tumor tissue sample available. Note: If the biopsy is considered by the investigator to pose an unacceptable safety risk to the patient or would compromise tumor measurements, the biopsy requirement may be waived for an individual patient after notification of the medical monitor. For patients without on-study screening biopsy, an archival FFPE tissue sample (block or 25 unstained slides) should be provided.
8. Adequate normal organ and marrow function as defined below:

   1. Absolute neutrophil count ≥ 1.5 x 109 cells/L
   2. Platelets ≥ 75 x 109/L
   3. Hemoglobin ≥ 8 g/dL
   4. Aspartate and alanine aminotransferases (AST, ALT) ≤ 3 x upper limit of normal (ULN) and alkaline phosphatase <2.5x ULN
   5. Thyroid stimulating hormone (TSH) within normal limits, or Total triiodothyronine (T3) is within normal limits, or Free T3 and free thyroxine (T4) are within the normal limits
   6. Total bilirubin ≤ 2 x ULN (except patients with documented Gilbert's syndrome; up to 3 x ULN)
   7. Creatinine < 2 mg/dl (or a glomerular filtration rate > 60)
9. Female patients of childbearing potential (WOCBP) must provide a negative urine pregnancy test 72 hours prior to the first administration of study treatment, and must agree to: (I) use a medically accepted and highly effective birth control method (i.e. those with a failure rate less than 1%; refer to Appendix 6); (II) refrain from donating ovules; and (III) refrain from breastfeeding for the duration of the study treatment and for 180 days after the last dose of cemiplimab.

   - A woman is considered of childbearing potential ( i.e. fertile) following menarche and until becoming postmenopausal unless permanently sterile. Women will be considered postmenopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:
   1. Amenorrheic for ≥1 year in the absence of chemotherapy and/or hormonal treatments
   2. Luteinizing hormone (LH) and/or follicle stimulating hormone and/or estradiol levels in the postmenopausal range
   3. Radiation induced oophorectomy with last menses >1 year ago
   4. Chemotherapy induced menopause with >1 year interval since last menses
   5. Surgical sterilization (bilateral oophorectomy or hysterectomy)
   6. Women <50 years of age would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
   7. Women ≥50 years of age would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
10. Male participants of reproductive potential are eligible to participate if they agree to the following starting with the first dose of study treatment through at least 180 days (a spermatogenesis cycle) after the last dose of study treatment:

    1. Refrain from donating sperm plus, either:
    2. Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent, or
    3. Must agree to use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception, as a condom may break or leak, when having sexual intercourse with a WOCBP who is not currently pregnant.

Exclusion Criteria:

1. Distant metastatic disease (M1), visceral and/or distant nodal.
2. Patients who have another malignancy that is progressing or requires active treatment, except:

   1. Non-melanoma skin cancer that has undergone potentially curative therapy In situ cervical carcinoma
   2. Any tumor that has been deemed to be effectively treated with definitive local control (with or without continued adjuvant hormonal therapy).
3. Patients who have received a previous systemic treatment for cancer within the last previous 3 months or 5 half-lives (whichever is latest), including immunotherapy, prior to initiation of dosing within this protocol.
4. History of, or significant evidence of risk for, severe chronic inflammatory or autoimmune disease.

   Note: Patients with vitiligo, type I diabetes mellitus, and endocrinopathies (including hypothyroidism due to autoimmune thyroiditis) only requiring hormone replacement, childhood asthma that has resolved, or psoriasis that does not require systemic treatment are permitted.
5. Patients who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load before randomization.

   Note: Patients should remain on antiviral therapy throughout trial treatment and follow.
6. Patients with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
7. Patients with known HIV who have controlled infection (undetectable viral load and CD4 count above 100 on a stable antiviral regimen) are permitted. For patients with controlled HIV infection, monitoring will be performed per local standards.
8. Active tuberculosis.
9. Receipt of a live vaccine within 28 days of enrollment.
10. Prior allogeneic stem cell transplantation, or autologous stem cell transplantation.
11. Recipient of a solid organ transplant (other than corneal transplants).
12. History of interstitial lung disease (eg, idiopathic pulmonary fibrosis, organizing pneumonia) or active, noninfectious pneumonitis that required immune-suppressive doses of glucocorticoids to assist with management.
13. Potential requirement for systemic corticosteroids or concurrent immunosuppressive drugs based on prior history or received systemic steroids within the last 2 weeks prior to enrollment.

    Notes: Physiologic replacement doses are allowed even if they are >10 mg of prednisone/day or equivalent. Inhaled or topical steroids at standard doses are allowed. Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication are eligible for the study.
14. Has participated in a study of an investigational agent or an investigational device within 4 weeks of enrollment.
15. Dementia or significantly altered mental status, or any social or economic conditions that would prohibit or interfere with the understanding or rendering of informed consent and compliance with the requirements of this protocol.
16. Female patients who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence adverse events (AE) and treatment-related AEs (TRAEs) assessed by NCI CTCAE v5.0 | During DLT evaluation period, the first 3 weeks of treatment for each patient
  The incidence of DLTs evaluated in Phase Ib: considered as the rate of patients who experience adverse events (AE) and treatment-related AEs (TRAEs) assessed by NCI CTCAE v5.0 which may be considered DLTs.
Relapse-Free Survival (RFS) rate at 3 years. | Throughout the study period, at 3 years from the start of treatment
  Relapse-Free Survival (RFS) rate at 3 years evaluated in Phase II study. 3-years RFS rate is defined as the percentage of patients free of locoregional progression or recurrence or new basocellular tumors, distant metastasis (RECIST v 1.1) or death due to any cause after 3 years from the date of study treatment. Patients not presenting any of the previous events will be censored at the date of last assessment. RFS will be summarized using the Kaplan-Meier method and displayed graphically where appropriate. The Cox proportional hazards model will be fitted to compute the hazard ratios on potential stratified groups if applicable. RFS will be calculated as median / mean (95% CI) for each cohort and RFS rate for different timepoints as applicable.The primary endpoint will be assessed locally and centrally. Central assessment will be prioritized for the primary endpoint.

SECONDARY OUTCOMES:
Pathological response assessment | Throughout the study period, at at 3 years from the start of treatment]
  Considered the proportion of patients with pathologic complete response (pCR) per Immune-Related Pathologic Response Criteria' (irPRC) criteria: considered as the rate of patients who achieve a pCR. The pCR rate will be estimated by binomial proportion, dividing the number of patients with pCR by the number of patients assessed. The primary analysis will be performed in the per protocol population to avoid missed patients who are not evaluable due to lost to follow up or other reasons. The corresponding exact 2-sided 95% CIs will be provided in global and by cohort..
Objective response rate (ORR) | Throughout the study period, at 3 years from the start of treatment
  Objective response rate (ORR) be considered as the percentage/proportion of patients with complete response (CR) or partial response (PR) as their overall best response throughout the study period. The ORR will be estimated by binomial proportion, dividing the number of patients with objective response (CR or PR). The corresponding exact 2-sided 95% CIs will be provided by cohort. Changes in tumor size from baseline will be calculated and displayed graphically, where appropriate.
Clinical benefit rate (CBR) | Throughout the study period, at at 3 years from the start of treatment
  Percentage/proportion of patients with complete response (CR) or partial response (PR), according to ORR definition for the trial, or maintained stable disease (SD) as their overall best response until surgery. The CBR will be estimated by binomial proportion, dividing the number of patients with objective response (CR, PR, or SD until surgery). The corresponding exact 2-sided 95% CIs will be provided by cohort. Changes in tumor size from baseline will be calculated and displayed graphically, where appropriate
Duration of clinical benefit (DBC) | Throughout the study period, at at 3 years from the start of treatment
  Defined as the time from first dose of treatment until relapse / progression or death from any cause, whichever occurs first, in patients who had a best overall response of CR, PR, or SD until surgery. Those patients without relapse /progression or death event will be censored on the date of their last tumor assessment. DCR will be summarized by cohort using Kaplan-Meier method and displayed graphically, where appropriate. The mean, median DCR and 95% CIs will be provided.
Rate of resectability, and downstaging: | Throughout the study period, at 6 months from the start of treatment
  defined as the percentage of patients who are eligible to surgical intervention after 4 cycles of neoadjuvant study treatment according to investigator criteria and achieve a complete resection (R0). Downstaging, defined as the percentage of patients that have a significant tumor decrease which would require a less complex surgical procedure and therefore less extensive functional and aesthetic consequences. The level of surgical complexity should be reduced to at least 1 lower level (for example, from a stage A surgical procedure to a stage B surgical procedure
Overall survival (OS) | Throughout the study period, at 3 years from the start of treatment
  Defined as the time from the date of study treatment initiation to the date of death for any cause. The follow-up of subjects still alive will be censored at the date of last visit/contact. OS will be summarized using the Kaplan-Meier method and displayed graphically where appropriate. CIs for the 25th, 50th and 75th percentiles or specific time points considered adequate by the time of the analysis will be reported. The Cox proportional hazards model will be fitted to compute the hazard ratios on potential stratified groups if applicable. OS will be calculated as median / mean (95% CI) for each cohort and OS rate for different timepoints as applicable.

CONTACTS AND LOCATIONS:
Overall Officials: María González Cao, M.D., Ph.D., Study Chair — Medical oncology Department / Dr Rosell Oncologic Institute. Hospital Dexeus, Barcelona, Spain; Susana Puig, M.D., Ph.D., Study Chair — Hospital Clinic of Barcelona
Locations (4):
- Spain (4):
  - Hospital Universitario Dexeus - Grupo Quirónsalud. Carrer de Sabino Arana, 19 Ed, Distrito de Les Corts, Barcelona, Barcelona
  - Hospital Clínic de Barcelona. Carrer de Villarroel, 170, L'Eixample, Barcelona, Barcelona
  - Hospital Ramón y Cajal. M-607, Km. 9, 100, Fuencarral-El Pardo,, Madrid, Madrid
  - Hospital Miguel Servet de Zaragoza. P.º de Isabel la Católica, 1-3, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No